CLINICAL TRIAL: NCT03957889
Title: Correlation Between Students' and Trainers' Evaluations While Learning Delegated Surgical Procedures: a Prospective Cohort Study
Brief Title: Students and Trainers' Evaluations Correlation
Status: Completed | Type: Observational
Sponsor: Centre de l'arthrose, Paris (Other)
Collaborators: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Principal Investigator, Maillot Cédric, MD, MSC, Centre de l'arthrose, Paris
Other Study IDs: nurse_pedago
Record Dates: First submitted 2019-05-19; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Surgical Procedure, Unspecified; Critical Thinking; Simulation; Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Student
  Interventions: Other: Educational simulation
- Trainers
  Interventions: Other: Educational simulation

INTERVENTIONS:
Other: Educational simulation

SUMMARY:
The delegation of procedures within the medical competence to the nurses can increase the effectiveness of the healthcare provided. The objectives of the study are (1) to assess the quality of training courses for delegated surgical procedures through implementation for graduate scrub nursing ("students") (2) and to evaluate the correlation between the evaluation of this training carried out by students and the self-assessment conducted by the faculty ("trainers").

ELIGIBILITY:
Inclusion Criteria:

* scrub nurses already in practice
* professional trainer, specialist in the field of the proposed course subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We divided Students into groups of 10 to 12 students, distributed into 5 sessions over the study period. We paid attention to mix these groups according to various places of exercise, surgical skills, length of professional practice and sectors of public or private activities. This group allocation was intended to enrich the exchanges between students by providing diverse personal and professional experiences, while maintaining a balance between the groups.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
SFDP26 questionnaire | 2 weeks
  This questionnaire is part of the System for Evaluation of Teaching Qualities (SETQ) which includes (1) a self-assessment by the trainer (2) an assessment by the student (3) then a feedback and (4) a follow-up to improve teaching. The SFDP26 questionnaire therefore exists in several versions for an evaluation of training by the students but also for a self-evaluation of by the trainers. Both versions share 25 basic items covering 7 dimensions of teaching quality

IPD SHARING:
Plan to Share IPD: No